CLINICAL TRIAL: NCT03248518
Title: Lessening the Impact of Fatigue in Inflammatory Rheumatic Diseases: A Randomised Clinical Trial
Brief Title: Lessening the Impact of Fatigue in Inflammatory Rheumatic Diseases
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Versus Arthritis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.049.16; Epi029 (Other: Epidemiology Group, University of Aberdeen)
Record Dates: First submitted 2017-02-15; First posted 2017-08-14 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis; Lupus Erythematosus, Systemic; Axial Spondyloarthritis; Psoriatic Arthritis; Sjogren's Syndrome
Keywords: Inflammatory Rheumatic Disease; Fatigue; Exercise; Behavioural Intervention; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Axial Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Axial Spondyloarthritis; Arthritis, Psoriatic; Sjogren's Syndrome; Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care alone (Active Comparator): Participants receive written information about fatigue which is designed as self-management guide.
  Interventions: Behavioral: Usual Care
- CBA + usual care (Active Comparator): In addition to usual care, participants receive a talking therapy using a cognitive behavioural approach. The talking therapy will be delivered via telephone by a trained rheumatology health care professional who will contact the participant for 8 sessions over a period of 6 months.
  Interventions: Behavioral: Usual Care; Behavioral: Cognitive behavioural approach
- PEP + usual care (Active Comparator): In addition to usual care, participants receive a personalised exercise programme. After an initial face-to-face assessment, the remaining programme will be delivered via telephone by a trained rheumatology health care professional who will contact the participant for 7 sessions over a period of 6 months.
  Interventions: Behavioral: Usual Care; Behavioral: Personalised Exercise Programme

INTERVENTIONS:
Behavioral: Usual Care — Information booklet on fatigue which represents usual care in almost all UK rheumatology centres
Behavioral: Cognitive behavioural approach — A talking therapy which explicitly aims to replace unhelpful beliefs and behaviours through the application of patient-centred strategies and behavioural activities
  Other Names: CBA
  Arms: CBA + usual care
Behavioral: Personalised Exercise Programme — PEP is a graded exposure behaviour therapy which aims to gradually optimise patients levels of physical activity with view to modifying their altered perception of effort and ultimately reduce the severity and impact of fatigue.
  Other Names: PEP
  Arms: PEP + usual care

SUMMARY:
Fatigue is common and disabling for most patients with inflammatory rheumatic disease. Therapies designed to improve physical activity and 'talking' treatments, which positively help patients change the way they think and behave, are both helpful in reducing the burden of the fatigue. However, few patients have access to these treatments in most health services. This situation results from the absence of standardised programmes and limited availability of relevant therapists.

The investigators aim to enhance access to fatigue alleviating physical activity and talking therapies by testing innovative,standardised and cost-effective approaches to treatment delivery.

The investigators will also use this opportunity to understand how to select the best treatment for a patient based on their individual profile and to better understand how these treatments actually work. This in turn may lead to more refined and effective therapies in the future.

DETAILED DESCRIPTION:
Eligible participants will be identified from patients with inflammatory rheumatic diseases attending major secondary care rheumatology services in the United Kingdom. Potential participants will be identified using local databases/clinic lists and will then be mailed a pre-study invite, which will include questions about fatigue. Potentially eligible participants will be invited to attend a baseline assessment.

Once it has been confirmed at the baseline assessement that they are eligible to take part in the study, the consented participant will be allocated to one of three treatment groups. During the course of the trial, the participant will be invited to visit the study centre three more times for assessments.

At each of the four assessment visits (baseline, and approximately 2, 7 and 13 months after) they will be asked:

1. To complete questionnaires which collect information about various outcomes which we think will improve in response to the therapies under evaluation as well as factors which will help us understand how the treatments may work, and factors which may help identify those patients better suited to one therapy over another
2. To provide a blood sample for research
3. To take part in an aerobic fitness test
4. To wear an activity monitor for the next 7 days which will be fitted at each visit
5. To answer three short questions about engagement with intervention delivered by telephone from trial office at the time of session 4 and 8 (CBA and PEP intervention only). Similarly, the allocated therapists will be asked to give their view of the participants' engagement with the intervention.

All participants will be asked to keep a diary on any other treatments they are using in addition to the treatments they may receive during the study and how costly these other treatments are. The diary period will last for the first 6 months and then for 2 weeks after the third visit and 2 weeks before the last visit.

After they finished the study, the investigators may approach a subgroup of participants who received either the talking therapy or the personalised exercise programme again and ask for an interview to enable more detailed feedback on if they found the intervention helpful and how it has changed their daily life.

ELIGIBILITY:
Inclusion Criteria:

* be ≥ 18 years at the time of consent
* have been diagnosed with rheumatoid arthritis (RA), systemic lupus erythematous (SLE), axial spondyloarthritis (AxSpA) or psoriatic arthritis (PSA) by a rheumatologist
* report fatigue to be a persistent problem
* have access to a telephone landline or mobile telephone and/or internet based audio/video calls
* give permission for researchers to access their hospital medical notes
* currently be under the care of a secondary care physician
* have stable disease as evidenced by no change in immunomodulatory therapy within the last three months based on the hospital medical record

Exclusion Criteria:

* there are significant abnormalities of thyroid function (TSH levels) on the most recent blood test done within the last three months
* there is evidence of severe anaemia (haemoglobin levels) on the most recent blood test done within the last three months
* there is evidence of severe renal dysfunction (eGFR) on the most recent blood test done within the last three months
* they have a medical condition which would make the proposed interventions unsuitable, e.g. significant heart disease
* they are pregnant
* they are unable to understand English sufficiently to take part in the intervention
* they are unable to provide written informed consent
* they are not willing to be randomised
* they are currently participating in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Fatigue (severity) using Chalder Fatigue Scale (Likert) | 56 weeks
  Chalder Fatigue Scale (Likert), assessed at 56 weeks after baseline, between-group change CBA+UC vs UC and PEP+UC vs UC with main estimate of treatment effect at 56 weeks after randomisation, Main estimate of treatment effect at 56 weeks
Fatigue (severity) using Chalder Fatigue Scale (Likert) | 10 weeks
  Chalder Fatigue Scale (Likert), assessed at 10 weeks after baseline, between-group change CBA+UC vs UC and PEP+UC vs UC
Fatigue (severity) using Chalder Fatigue Scale (Likert) | 28 weeks
  Chalder Fatigue Scale (Likert), assessed at 28 weeks after baseline, between-group change CBA+UC vs UC and PEP+UC vs UC
Fatigue (impact) using Fatigue Severity Scale | 56 weeks
  Fatigue Severity Scale, co-primary outcome assessed at 56 weeks after baseline, between-group change CBA+UC vs UC and PEP+UC vs UC with main estimate of treatment effect at 56 weeks
Fatigue (impact) using Fatigue Severity Scale | 10 weeks
  Fatigue Severity Scale, co-primary outcome assessed at 10 weeks after baseline, between-group change CBA+UC vs UC and PEP+UC vs UC
Fatigue (impact) using Fatigue Severity Scale | 28 weeks
  Fatigue Severity Scale, co-primary outcome assessed at 28 weeks after baseline, between-group change CBA+UC vs UC and PEP+UC vs UC

SECONDARY OUTCOMES:
Fatigue (physical, living, cognition and emotional aspects) using Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire | 0, 10 weeks, 28 weeks, 56 weeks after randomisation
  Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire
Quality of life & health utility index | 0, 10 weeks, 28 weeks, 56 weeks after randomisation
  SF-12
Pain using numerical rating scale | 0, 10 weeks, 28 weeks, 56 weeks after randomisation
  Pain numerical rating scale
Anxiety and depression using Hospital anxiety and depression scale | 0, 10 weeks, 28 weeks, 56 weeks after randomisation
  Hospital anxiety and depression scale
Impact on work using Work Productivity and Activity Impairment Questionnaire | 0, 10 weeks, 28 weeks, 56 weeks after randomisation
  Work Productivity and Activity Impairment Questionnaire: Specific Health Problem
Impact on activities using Valued Life Activities Scale | 0, 10 weeks, 28 weeks, 56 weeks after randomisation
  Valued Life Activities Scale
Change of global health | 10 weeks, 28 weeks, 56 weeks after randomisation
  Single question to indicate perceived change in global health compared with last assessment visit

CONTACTS AND LOCATIONS:
Overall Officials: Gary Macfarlane, PhD, Principal Investigator — University of Aberdeen; Neil Basu, MBChB, PhD, Principal Investigator — University of Glasgow
Locations (6):
- United Kingdom (6):
  - NHS Grampian, Aberdeen
  - NHS Tayside, Dundee
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Midlands Partnership NHS Foundation Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gray SR, Montoye AHK, Vondrasek JD, Neph S, Siebert S, Paul L, Bachmair EM, Basu N. Associations of physical activity levels with fatigue in people with inflammatory rheumatic diseases in the LIFT trial. Rheumatol Adv Pract. 2024 Aug 24;8(3):rkae106. doi: 10.1093/rap/rkae106. eCollection 2024. PMID 39257857
- [Derived] Bachmair EM, Martin K, Aucott L, Dhaun N, Dures E, Emsley R, Gray SR, Kidd E, Kumar V, Lovell K, MacLennan G, McNamee P, Norrie J, Paul L, Packham J, Ralston SH, Siebert S, Wearden A, Macfarlane G, Basu N; LIFT study group. Remotely delivered cognitive behavioural and personalised exercise interventions for fatigue severity and impact in inflammatory rheumatic diseases (LIFT): a multicentre, randomised, controlled, open-label, parallel-group trial. Lancet Rheumatol. 2022 Jun 27;4(8):e534-e545. doi: 10.1016/S2665-9913(22)00156-4. eCollection 2022 Aug. PMID 36388001
- [Derived] Martin KR, Bachmair EM, Aucott L, Dures E, Emsley R, Gray SR, Hewlett S, Kumar V, Lovell K, Macfarlane GJ, MacLennan G, McNamee P, Norrie J, Paul L, Ralston S, Siebert S, Wearden A, White PD, Basu N. Protocol for a multicentre randomised controlled parallel-group trial to compare the effectiveness of remotely delivered cognitive-behavioural and graded exercise interventions with usual care alone to lessen the impact of fatigue in inflammatory rheumatic diseases (LIFT). BMJ Open. 2019 Jan 30;9(1):e026793. doi: 10.1136/bmjopen-2018-026793. PMID 30705244
- See also: Click here for more information about this study — https://w3.abdn.ac.uk/hsru/lift/

DOCUMENTS (3):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03248518/Prot_001.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03248518/SAP_002.pdf
  • Informed Consent Form (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT03248518/ICF_003.pdf